CLINICAL TRIAL: NCT06628778
Title: Collaborative Risk-stratified Investigation in Teen Inpatients With Critical Illness: Anticoagulation With LMWH in Kids for ThromboProphylaxis (CRITICAL-Kids-TP)
Acronym: CRITICALKidsTP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00469377 - CRITICAL-Kids-TP
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism (VTE)
Keywords: pediatric; adolescent; critical illness; thromboprophylaxis
MeSH Terms: conditions — Venous Thromboembolism; Critical Illness | interventions — Dalteparin

STUDY DESIGN:
Intervention Model Description: PROBE study design, Randomized allocation 2:1 (Intervention:Standard of care) of dalteparin thromboprophylaxis versus standard-of-care (i.e., no pharmacological thromboprophylaxis). Analytic study populations will be modified intent-to-treat, per-protocol, and safety populations
Who Masked: Outcomes Assessor
Masking Description: Prospective Randomized Open, Blinded-Endpoint study design. There will be a blinded end-point adjudication committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dalteparin Thromboprophylaxis (Experimental): This arm will receive the study intervention, dalteparin thromboprophylaxis during pediatric intensive care unit hospitalization
  Interventions: Drug: Dalteparin
- Standard-of-Care Arm (No Intervention): This arm will receive standard of care (i.e., no pharmacological thromboprophylaxis)

INTERVENTIONS:
Drug: Dalteparin — Dalteparin thromboprophylaxis administered subcutaneously twice daily (every 12 hours) from enrollment through pediatric intensive care unit discharge
  Arms: Dalteparin Thromboprophylaxis

SUMMARY:
Critically ill adolescents are at greatest risk for developing hospital-acquired venous thromboembolism. To date, no phase 3 randomized controlled trials have been conducted for pharmacological thromboprophylaxis as primary venous thromboembolism prevention in children. The investigators will perform a United States definitive multicenter phase 3 randomized controlled trial of the low molecular weight heparin dalteparin as primary venous thromboembolism prophylaxis among critically ill adolescents who are classified a priori as high risk based upon the investigators validated risk prediction models.

DETAILED DESCRIPTION:
This trial will establish definitive evidence on the comparative efficacy and safety of pharmacological thromboprophylaxis with the low molecular weight heparin (LMWH) dalteparin versus standard of care (no pharmacological thromboprophylaxis) for the primary prevention of venous thromboembolism (VTE), including deep vein thrombosis and/or pulmonary embolism) among critically ill adolescents who meet a priori criteria for high risk of hospital-acquired (HA-) VTE. No anticoagulant has been FDA-approved for primary VTE prevention in hospitalized children. In the past two decades, the diagnosis of pediatric hospital-acquired VTE (HA-VTE) in the U.S. has increased 130-200-fold. The investigators have shown that critically-ill adolescents are one the highest risk subpopulations for HA-VTE, with average occurrence rates of 13.2% (range: 6.3-19.8%), and have derived and prospectively validated risk models for HA-VTE in this population. Despite a simultaneously increased risk of bleeding in critically ill adolescents, particularly after surgery or major trauma, an investigator-initiated multicenter phase 2 trial recently led by the investigators group during the COVID-19 pandemic demonstrated the safety of LMWH for primary HA-VTE prevention. To date, risk-stratified phase 3 Randomized Controlled Trials (RCTs) of LMWH thromboprophylaxis as primary HA-VTE prevention in children have not been performed. The investigators will perform a U.S.-based definitive multicenter phase 3 RCT of the LMWH dalteparin versus standard-of-care (SOC), no pharmacological thromboprophylaxis) for VTE prevention among critically ill adolescents at highest a priori risk for HA-VTE applying evidence from the investigators published risk prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Admission Age between 12- 18 years of age
* Within 24 hours of pediatric intensive care unit (PICU) admission for enrollment
* Presence of a Central Venous Catheter
* Anticipated PICU Length of Stay /= 4 days
* Presumed or confirmed infection or inflammatory condition

Exclusion Criteria:

* Active treatment for VTE or known VTE present prior to or on pediatric intensive care unit (PICU) admission
* Current receipt of an antithrombotic agent excluding unfractionated heparin for vascular catheter patency
* Active ISTH-defined clinically relevant bleeding
* Surgery in the last 7-days
* Major trauma within the last 7-days
* Admission for management of congenital heart disease including perioperative management of critical congenital heart disease
* Presence of coagulopathy including:
* International normalized ratio (INR) 2.0 activated partial thromboplastin time (aPTT) 50 seconds Platelet count 50 x103/mL
* Creatinine clearance 30 ml/min/1.73 m2
* Known hypersensitivity to heparin or pork products
* Laboratory confirmed heparin induced thrombocytopenia
* Current pregnancy or lactation,
* Presence of an epidural catheter
* Prior enrollment in the CRITICAL-Kids-TP Trial

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 802 (Estimated)
Dates: Start 2026-10-31 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Risk (i.e., cumulative incidence) of Symptomatic venous thromboembolism | From randomization through discharge from the pediatric intensive care unit, approximately 1-2 weeks
  International Society on Thrombosis and Haemostasis (ISTH) defined symptomatic venous thromboembolism
Risk (i.e., cumulative incidence) of Clinically relevant bleeding | From randomization through discharge from the pediatric intensive care unit, approximately 1-2 weeks
  International Society on Thrombosis and Haemostasis (ISTH) defined clinically relevant bleeding (Major bleeding + Clinically relevant Non-major bleeding)

SECONDARY OUTCOMES:
Net Clinical Benefit - Modelled Attributable Risk Difference in HA-VTE (Efficacy) by Attributable Risk Difference in clinically relevant bleeding (Safety) | From randomization through discharge from the pediatric intensive care unit, approximately 1-2 weeks
  Net clinical benefit is a bivariate endpoint analysis (i.e., trade-off between venous thromboembolism and bleeding risks as described below). One-year risks and corresponding 95% confidence intervals (CI) of hospital-acquired venous thromboembolism and clinically relevant bleeding for each study arm will be calculated from weighted Kaplan-Meier curves. A bivariate decision curve will be specified using the 12-month absolute risk difference for venous thromboembolism and bleeding outcomes. The bivariate outcomes for dalteparin and standard-of-care arms will be compared under a hypothesis of superiority using the superiority boundary of a bivariate endpoint analysis, with inference based on the 95% confidence rectangle (i.e., the rectangle defined by the 95% CI for hospital-acquired venous thromboembolism absolute risk difference and the 95% CI for bleeding absolute risk difference). Superiority will be decided if the 95% confidence rectangle rules out the superiority curve.
Risk (i.e. cumulative incidence) of symptomatic venous thromboembolism | From randomization through 30-days post discharge from the pediatric intensive care unit
  International Society on Thrombosis and Haemostasis-defined symptomatic venous thromboembolism
Risk (i.e. cumulative incidence) of clinically relevant bleeding | From randomization through 30-days post discharge from the pediatric intensive care unit
  International Society on Thrombosis and Haemostasis-defined clinically relevant bleeding (Major Bleeding + Clinically Relevant Non-Major Bleeding)
Serious adverse events | From randomization through 30-days post discharge from the pediatric intensive care unit
  As federally defined.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sochet, MD, MSc, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children"s Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Sochet AA, Amankwah EK, Andalib V, Jaffray J, Male C, Faustino EV, Goldenberg NA; Pedi-ATLAS Group and the Antithrombotic Trials Working Party of the Pediatric Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Enhanced trial efficiency of the novel "contemporaneous control recapture" parallel-cohort RCT design: Methods and application in the CRITICAL-Kids-TP trial. Contemp Clin Trials. 2026 Jan;160:108142. doi: 10.1016/j.cct.2025.108142. Epub 2025 Nov 10. PMID 41223938